CLINICAL TRIAL: NCT04751773
Title: Postoperative Exercise Training in Patients With Colorectal Liver Metastases Undergoing Surgery (ELMA)
Acronym: ELMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jesper Frank Christensen, PhD, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELMA
Record Dates: First submitted 2021-01-29; First posted 2021-02-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Liver Metastasis
Keywords: Aerobic exercise; Resistance exercise; Perioperative medicine; Prehabilitation; Rehabilitation; Cancer; Surgical oncology; Surgery; Exercise oncology
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants and the exercise intervention instructors cannot be blinded, given the nature of the intervention. The outcome assessors of the primary and key secondary outcomes (adverse events and markers of surgical stress, respectively) will be blinded. For practical reasons, the outcome assessors of the following secondary outcomes will be not be blinded: resting cardiovascular factors, aerobic capacity, muscle strength, functional performance, and body composition and anthropometrics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care alone (CON) (No Intervention): Participants allocated to CON receive the standard patient care program, as provided by Rigshospitalet, Copenhagen, Denmark.
  Participants allocated to CON are allowed to exercise on their own initiative or participate in any standard care hospital- or municipality-based exercise training program.
- Postoperative exercise training and standard care (EX) (Experimental): Participants allocated to EX receive the standard patient care program, as provided by Rigshospitalet, Copenhagen, Denmark, and postoperative exercise training.
  The postoperative exercise training program consists of 8 weeks of supervised and home-based exercise 5 times/week. The intensity and duration are progressively increased during the postoperative period
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Perioperative exercise training
  Arms: Postoperative exercise training and standard care (EX)

SUMMARY:
Surgery is a primary treatment modality in the intended curative treatment of colorectal liver metastases (CRLM). However, surgery elicits a cascade of potentially detrimental stress responses that may drive the onset of long-term disease progression. Exercise training is emerging as an adjunct treatment in surgical oncology and holds potential to modify the surgical stress response. Against this background, we designed the present randomized controlled trial to evaluate the therapeutic role of pre- and postoperative exercise training in patients with CRLM undergoing open liver resection.

DETAILED DESCRIPTION:
BACKGROUND:

Colorectal cancer is the third most frequent type of cancer in Denmark, with more than 5000 new cases annually. Colorectal liver metastases (CRLM) develop in nearly one fourth of all patients with colorectal cancer, and poses a poor prognostic outlook, with low survival rates and short time to disease progression. Surgical resection, either upfront or following downstaging with perioperative treatments, confers substantial survival benefit in patients with CRLM, and may even comprise a curative treatment modality. However, surgery elicits a cascade of biological responses characterized by increased dissemination of tumor cells and modulation of neuroendocrine, inflammatory, and immunological factors. These local and systemic perturbations typically persist for days to weeks following surgery and may independently or in concert drive the onset of long-term disease progression. Under normal physiological conditions, exercise training is a potent modulator of immune function, systemic inflammation, and the neuroendocrine system, raising the possibility that perioperative exercise training may ameliorate the surgical stress response during and after surgery. However, in a recent systematic review and meta-analysis (submitted), we found that the effects and safety of preoperative and early postoperative exercise are unknown in patients with gastrointestinal cancers (including CRLM) due to lack of studies, widespread methodological issues, and poor ascertainment and reporting of adverse events. Safety is arguably the single most important consideration for the application perioperative exercise, and methodological robust trials evaluating the safety and tolerability of perioperative exercise training along with preliminary information on treatment efficacy are needed to inform the application of exercise in surgical oncology.

Against this background, we designed the present randomized controlled trial to evaluate the therapeutic role of postoperative exercise training in patients with CRLM undergoing open liver resection. The primary trial objective and hypothesis are:

1. To compare the number of serious adverse events (SAE) in standard care plus postoperative exercise (EX) vs. standard care alone (CON) in patients with colorectal liver metastases scheduled to undergo open liver resection. The primary research hypothesis is that the number of SAEs is non-inferior in EX vs. CON

   The key secondary study objectives and hypotheses are:
2. To compare the effect of EX vs. CON on incidence of postoperative hospital admissions in patients with CRLM undergoing surgery. We hypothesize that the incidence of postoperative hospital admissions are non-inferior in EX vs. CON
3. To compare the effect of EX vs. CON on relative dose intensity of adjuvant chemotherapy and time from surgery to initiation of adjuvant chemotherapy in patients with CRLM undergoing surgery. We hypothesize that the relative dose intensity of adjuvant chemotherapy and time from surgery to initiation of adjuvant chemotherapy are non-inferior in EX vs. CON.
4. To compare the effect of EX vs. CON on selected patient-reported symptomatic adverse events in patients with CRLM undergoing surgery
5. To compare the effect of EX vs. CON on surgical stress responses (neuroendocrine, inflammatory, and immune factors) in patients with CRLM undergoing surgery.

   The secondary study objectives are:
6. To evaluate the feasibility of EX.
7. To compare the effect of EX vs. CON on functional capacity, muscle strength, aerobic capacity, and body composition in patients with CRLM undergoing surgery.
8. To compare the effect of EX vs. CON on clinical outcomes in patients with CRLM undergoing surgery.
9. To compare the effect of EX vs. CON on patient-reported outcomes in patients with CRLM undergoing surgery.
10. To compare the effect of EX vs. CON on circulating tumor DNA and DNA methylation in patients with CRLM undergoing surgery
11. To evaluate the effects of acute pre- and postoperative exercise on neuroendocrine, immunological, and inflammatory factors in patients with CRLM undergoing surgery.
12. To conduct explorative preclinical sub-studies.

TRIAL DESIGN:

This trial is a single-center, randomized, controlled, parallel-group trial performed at Centre for physical Activity (CFAS), Rigshospitalet, Copenhagen, Denmark, and Department of Surgical Gastroenterology, Rigshospitalet, Copenhagen, Denmark.

A total of 60 participants with CRLM will be included and randomly allocated 2:1 to standard care and postoperative exercise training (EX) or standard care alone (CON). The participants will undergo two trial visits at CFAS during the study period: One preoperative trial visit (1-3 days after inclusion and 2-7 days before surgery) and one post-surgery trial visit (8 weeks after discharge). For each visit, the participants will be assessed for body composition and anthropometrics, resting cardiovascular factors, standard blood biochemistry, aerobic capacity (VO2peak, ventilatory threshold), maximal muscle strength, and functional performance. In addition, blood samples will be taken before, during, and immediately after surgery, and on post-operative day 1, 3, and 15 and neuroendocrine, inflammatory, and immune factor will be analyzed. Patient-reported outcomes will be collected at all trial visits and 1, 2, and 3 years after randomization. Data from medical records regarding mortality and disease recurrence will be collected up to 3 years after randomization. As an optional procedure, we will collect blood samples before, during, and after a pre- and a postoperative supervised exercise training session.

ELIGIBILITY:
Inclusion Criteria: Participants diagnosed with colorectal liver metastasis planned for open surgery of liver metastases

Exclusion Criteria:

* Age <18
* Pregnancy
* Other known malignancy requiring active cancer treatment that prohibits execution of test or training procedures
* Conditions that prohibit execution of trial procedures
* Inability to understand the Danish language.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | From discharge to 8 weeks after discharge

SECONDARY OUTCOMES:
Postoperative hospital admissions | From discharge to 8 weeks after discharge
  Incidence of postoperative hospital re-admissions, defined as any non-scheduled ≥ 24 h hospitalization
Relative dose intensity (RDI) of adjuvant chemotherapy | From date of planned initiation of adjuvant chemotherapy until 8 weeks after discharge
  RDI (%) of adjuvant chemotherapy, calculated as the actual dose intensity / standard dose intensity x 100%
Time to initiation of adjuvant chemotherapy | From surgery until 8 weeks after discharge
  Time from surgery to initiation of adjuvant chemotherapy
Patient-reported symptomatic adverse events | Baseline, 7 days after discharge, 7 days after each administration of adjuvant chemotherapy, 8 weeks after discharge.
  Patient-reported symptomatic adverse events, assessed using the using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Surgical stress: IL-1β | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood IL-1β concentration
Surgical stress: IL-6 | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood IL-6 concentration
Surgical stress: IL-8 | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood IL-8 concentration
Surgical stress: IL-10 | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood IL-10 concentration
Surgical stress: interferon- γ | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood interferon- γ concentration
Surgical stress: C-reactive protein | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood C-reactive protein
Surgical stress: Leukocyte differential counts | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood leukocyte cell counts (total and per type [eosinophils, basophils, lymphocytes, monocytes, neutrophils])
Surgical stress: Natural killer (NK) cells | Baseline, after resection, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood NK cell count
Surgical stress: T cells | Baseline, after resection, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood T cell count
Surgical stress: Adrenocorticotropic hormone (ACTH) | After last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 15
  Changes in blood ACTH concentration
Surgical stress: Cortisol | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood cortisol concentration
Surgical stress: Adrenaline | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood adrenaline concentration
Surgical stress: Noradrenaline | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in blood noradrenaline concentration

OTHER OUTCOMES:
3-years cancer-specific survival | Randomization to 3 years after randomization
  Proportion of patients who have not died from colorectal cancer 3 years after randomization
3-years overall survival | Randomization to 3 years after randomization
  Proportion of patients who are alive 3 years after randomization
Carcinoembryonic antigen (CEA) | Baseline, postoperative day 15, 8 weeks after discharge
  Changes in blood CEA
Circulating tumor DNA (ctDNA) | Baseline, postoperative day 15, 8 weeks after discharge
  Changes in blood ctDNA
DNA methylation | Baseline, 3 days before surgery, 1 h before anesthesia, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in DNA methylation
Exercise feasibility: Exercise sessions attendance rate | From baseline to 8 weeks after discharge
  Exercise sessions attendance rate (%), defined as number of attended exercise sessions / number of prescribed exercise sessions x 100
Exercise feasibility: Relative dose intensity (RDI) of exercise | From baseline to 8 weeks after discharge
  RDI (%) of exercise, defined as prescribed exercise dose / performed exercise dose x 100
Exercise feasibility: Early termination of exercise sessions | From baseline to 8 weeks after discharge
  Incidence of early termination of attended exercise sessions, defined as termination of an exercise session before the prescribed exercises have been performed
Exercise feasibility: Exercise intervention interruptions | From baseline to 8 weeks after discharge
  Incidence of exercise intervention disruptions, defined as a period of ≥ 7 days without an attended exercise session
Exercise feasibility: Exercise sessions requiring dose modifications | From baseline to 8 weeks after discharge
  Incidence of exercise sessions requiring dose modifications, defined as any deviation from the prescribed exercise
Exercise feasibility: Permanent discontinuation of the exercise intervention | From baseline to 8 weeks after discharge
  Incidence of permanent discontinuations of the exercise intervention, defined as participants that withdraw entirely from the exercise intervention, regardless of whether they remain in the trial
Exercise feasibility: Time from discharge to initiation of postoperative exercise | From surgery to 8 weeks after discharge
  Time from discharge to first attended postoperative exercise session
Exercise feasibility: Patient-reported symptomatic adverse events (paint, dizziness, nausea, fatigue, other) | Immediately before and immediately after each exercise session performed from baseline to 8 weeks after discharge
  Changes in patient-reported symptomatic adverse events (paint, dizziness, nausea, fatigue, other)
Intraoperative factors: Blood loss during surgery | During surgery
  Blood loss during surgery
Intraoperative factors: Duration of surgery | During surgery
  Duration of surgery
Intraoperative factors: Blood transfusions | During surgery
  Incidence of blood transfusions
Resting cardiovascular factors: Resting systolic blood pressure | Baseline, 8 weeks after discharge
  Changes in resting systolic blood pressure
Resting cardiovascular factors: Resting diastolic blood pressure | Baseline, 8 weeks after discharge
  Changes in resting diastolic blood pressure
Resting cardiovascular factors: Resting heart rate | Baseline, 8 weeks after discharge
  Changes in resting heart rate
Resting cardiovascular factors: Hemoglobin concentration | Baseline, after last incision, after resection, 3 hour post-surgery, postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in hemoglobin concentration
Aerobic capacity: Peak oxygen consumption | Baseline, 8 weeks after discharge
  Changes in peak oxygen consumption assessed during an incremental exercise test (ergometer bicycling) to volitional exhaustion
Aerobic capacity: Ventilatory threshold | Baseline, 8 weeks after discharge
  Changes in ventilatory threshold assessed during an incremental exercise test (ergometer bicycling) to volitional exhaustion
Aerobic capacity: Peak power output | Baseline, 8 weeks after discharge
  Changes in peak power output assessed during an incremental exercise test (ergometer bicycling) to volitional exhaustion
Muscle strength: Leg press maximal muscle strength | Baseline, 8 weeks after discharge
  Changes in leg press one repetition maximum (1RM)
Muscle strength: Chest press muscle strength | Baseline, 8 weeks after discharge
  Changes in chest press 1RM
Muscle strength: Hand grip strength | Baseline, 8 weeks after discharge
  Changes in hand grip strength, assessed using a dynamometer
Functional performance: Habitual gait speed | Baseline, 8 weeks after discharge
  Changes in habitual gait speed
Functional performance: Maximal gait speed | Baseline, 8 weeks after discharge
  Changes in maximal gait speed
Functional performance: Stair climbing power | Baseline, 8 weeks after discharge
  Changes in stair climbing power
Body composition and anthropometrics: Body mass | Baseline, 8 weeks after discharge
  Changes in body mass
Body composition and anthropometrics: Body mass index | Baseline, 8 weeks after discharge
  Changes in body mass index
Body composition and anthropometrics: Total lean mass | Baseline, 8 weeks after discharge
  Changes in total lean mass, assessed by dual energy x-ray absorptiometry (DXA)
Body composition and anthropometrics: Appendicular lean mass | Baseline, 8 weeks after discharge
  Changes in appendicular lean mass, assessed by DXA
Body composition and anthropometrics: Abdominal fat mass | Baseline, 8 weeks after discharge
  Changes in abdominal fat mass, assessed by DXA
Body composition and anthropometrics: Total fat mass | Baseline, 8 weeks after discharge
  Changes in total fat mass, assessed by DXA
Body composition and anthropometrics: Fat percentage | Baseline, 8 weeks after discharge
  Changes in fat percentage, assessed by DXA
Body composition and anthropometrics: Hip circumference | Baseline, 8 weeks after discharge
  Changes in hip circumference
Body composition and anthropometrics: Waist circumference | Baseline, 8 weeks after discharge
  Changes in waist circumference
Standard blood biochemistry: Total cholesterol | Baseline, 8 weeks after discharge
  Changes in total cholesterol concentration
Standard blood biochemistry: Low-density lipoprotein cholesterol | Baseline, 8 weeks after discharge
  Changes in low-density lipoprotein cholesterol concentration
Standard blood biochemistry: High-density lipoprotein cholesterol | Baseline, 8 weeks after discharge
  Changes in high-density lipoprotein cholesterol concentration
Standard blood biochemistry: Triglyceride | Baseline, 8 weeks after discharge
  Changes in triglyceride concentration
Standard blood biochemistry: Glycated hemoglobin A1c | Baseline, 8 weeks after discharge
  Change in glycated hemoglobin A1c concentration
Standard blood biochemistry: Insulin | Baseline, 8 weeks after discharge
  Changes in insulin concentration
Standard blood biochemistry: Glucose | Baseline, 8 weeks after discharge
  Changes in blood glucose concentration
Health-related quality of life: Physical well-being | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported physical well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C)
Health-related quality of life: Social well-being | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported social well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C)
Health-related quality of life: Emotional well-being | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported emotional well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Health-related quality of life: Functional well-being | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported functional well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Health-related quality of life: Colorectal-cancer specific | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported colorectal-cancer specific health-related quality of life assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Health-related quality of life: General | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported general health-related qualify of life assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Health-related quality of life: Trial outcome index | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported trial outcome index assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Health-related quality of life: Total score (Functional Assessment of Cancer Therapy - Colorectal) | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported in health-related quality of life (total score) assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C).
Depression | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported depression, assessed using the Hospital Anxiety and Depression Scale (HADS).
Anxiety | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported anxiety, assessed using the Hospital Anxiety and Depression Scale (HADS).
Self-reported physical activity: Walking | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported weekly duration of walking, assessed using the International Physical Activity Questionnaire (IPAQ)
Self-reported physical activity: Moderate intensity physical activity (PA) | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported weekly duration of moderate intensity PA, assessed using the International Physical Activity Questionnaire (IPAQ)
Self-reported physical activity: Vigorous intensity physical activity (PA) | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported weekly duration of vigorous intensity PA, assessed using the International Physical Activity Questionnaire (IPAQ)
Self-reported physical activity: Total physical activity (PA) | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported weekly duration of total PA, assessed using the International Physical Activity Questionnaire (IPAQ)
Self-reported physical activity: Sitting time | Baseline, 8 weeks after discharge, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Changes in patient-reported weekly sitting time, assessed using the International Physical Activity Questionnaire (IPAQ)
Effect of acute perioperative exercise: IL-1β | 10 min before exercise, immediately after aerobic exercise
  Changes in blood IL-1β concentration during acute perioperative exercise
Effect of acute perioperative exercise: IL-6 | 10 min before exercise, immediately after aerobic exercise
  Changes in blood IL-6 concentration during acute perioperative exercise
Effect of acute perioperative exercise: IL-8 | 10 min before exercise, immediately after aerobic exercise
  Changes in blood IL-8 concentration during acute perioperative exercise
Effect of acute perioperative exercise: IL-10 | 10 min before exercise, immediately after aerobic exercise
  Changes in blood IL-10 concentration during acute perioperative exercise
Effect of acute perioperative exercise: Interferon- γ | 10 min before exercise, immediately after aerobic exercise
  Changes in blood interferon- γ concentration during acute perioperative exercise
Effect of acute perioperative exercise: C-reactive protein | 10 min before exercise, immediately after aerobic exercise
  Changes in blood C-reactive protein concentration during acute perioperative exercise
Effect of acute perioperative exercise: Leukocyte differential counts | 10 min before exercise, immediately after aerobic exercise
  Changes in blood leukocyte cell counts (total and per type [eosinophils, basophils, lymphocytes, monocytes, neutrophils]) during acute perioperative exercise
Effect of acute perioperative exercise: Natural killer cells | 10 min before exercise, immediately after aerobic exercise
  Changes in blood natural killer cell count during acute perioperative exercise
Effect of acute perioperative exercise: T cells | 10 min before exercise, immediately after aerobic exercise
  Changes in blood T cell count during acute perioperative exercise
Effect of acute perioperative exercise: Adrenocorticotropic hormone (ACTH) | 10 min before exercise, immediately after aerobic exercise
  Changes in blood ACTH concentration during acute perioperative exercise
Effect of acute perioperative exercise: Cortisol | 10 min before exercise, immediately after aerobic exercise
  Changes in blood cortisol concentration during acute perioperative exercise
Effect of acute perioperative exercise: Adrenaline | 10 min before exercise, immediately after aerobic exercise
  Changes in blood adrenaline concentration during acute perioperative exercise
Effect of acute perioperative exercise: Noradrenaline | 10 min before exercise, immediately after aerobic exercise
  Changes in blood noradrenaline concentration during acute perioperative exercise
LPS-induced IL-6 production of whole blood | Baseline, after resection, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in concentation of IL-6 in LPS-stumulated whole blood
LPS-induced TNF-a production of whole blood | Baseline, after resection, postoperative day 1, postoperative day 3, postoperative day 15, 8 weeks after discharge
  Changes in concentation of TNF-a in LPS-stumulated whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Jesper F Christensen, PhD, Principal Investigator — Centre for Physical Activity Research, Rigshospitalet, University of Copenhagen, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomsen SN, Krabek R, Yfanti C, Sjoberg S, Sundberg A, Dalsgaard DM, Thomsen LM, Aasvang EK, Qvortrup C, Mau-Sorensen M, Pedersen BK, Larsen PN, Sillesen MH, Schultz NA, Christensen JF, Simonsen C. Postoperative Exercise Training in Patients with Colorectal Liver Metastases A Randomized Controlled Trial. Ann Surg. 2024 Nov 11. doi: 10.1097/SLA.0000000000006587. Online ahead of print. PMID 39523954